CLINICAL TRIAL: NCT07037056
Title: The Effects of Posture Correction Exercises and Soft Tissue Mobilization on Reducing Shoulder and Neck Pain in Breastfeeding Mothers
Brief Title: The Effects of Posture CS and STM on Reducing Shoulder and Neck Pain in Breastfeeding Mothers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall20/1003
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Shoulder Pain; Neck Pain
MeSH Terms: conditions — Shoulder Pain; Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shoulder and Neck Strengthening + Postural Correction Exercises (Experimental)
  Interventions: Combination Product: Shoulder and Neck Strengthening + Postural Correction Exercises
- Shoulder and Neck Strengthening + soft tissue mobilization (Active Comparator)
  Interventions: Combination Product: Shoulder and Neck Strengthening + soft tissue mobilization

INTERVENTIONS:
Combination Product: Shoulder and Neck Strengthening + Postural Correction Exercises — Physiotherapy exercises of Shoulder and Neck Strengthening + Postural Correction Exercises for shoulder and neck pain
  Arms: Shoulder and Neck Strengthening + Postural Correction Exercises
Combination Product: Shoulder and Neck Strengthening + soft tissue mobilization — Physiotherapy exercises of Shoulder and Neck Strengthening + soft tissue mobilization Exercises for shoulder and neck pain
  Arms: Shoulder and Neck Strengthening + soft tissue mobilization

SUMMARY:
Breastfeeding, though essential for the nourishment and development of newborns, often imposes significant musculoskeletal strain on mothers, particularly in the neck and shoulder regions. Prolonged static postures, repetitive feeding routines, and improper ergonomic positions contribute to mechanical stress, leading to chronic discomfort or pain during the postpartum period Postnatal women frequently assume awkward positions while nursing, such as forward head posture, rounded shoulders, and spinal flexion, which contribute to musculoskeletal dysfunctions . The cumulative load on the musculoskeletal and fascial systems during breastfeeding leads to muscle imbalances, myofascial tightness, and trigger point development.

DETAILED DESCRIPTION:
Current physiotherapy interventions emphasize posture education, ergonomic training, and targeted exercises to mitigate this pain. Posture correction exercises aim to improve alignment, decrease strain on muscles and joints, and enhance motor control in the upper quarter . Soft tissue moblization a manual therapy technique targeting fascial layers, has also shown promising results in improving mobility, reducing trigger point activity, and decreasing referred pain.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum period of up to 12 months

Exclusion Criteria:

* History of trauma or cervical disc pathology
* Neurological disorders
* Previous musculoskeletal surgeries

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 6 Month
  The Numeric Pain Rating Scale (NPRS) is an 11-point scale used to measure pain intensity, ranging from 0 (no pain) to 10 (worst pain imaginable).
Neck Disability Index (NDI) | 6 Months
  The Neck Disability Index (NDI) is a questionnaire used to assess how neck pain affects a person's daily life and disability. It consists of 10 items, each scored on a 0-5 scale, resulting in a total score ranging from 0 to 50. A higher score indicates greater perceived disability due to neck pain
Breastfeeding self efficacy scale | 6 months
  All items are preceded by the phrase ''I can always'' and rated on a 5-point Likert scale, ranging from 1 (not at all confident) to 5 (always confident). Total scores range from 14 to 70, with higher scores reflecting more significant levels of breastfeeding self-efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Lahore City, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No